CLINICAL TRIAL: NCT02549313
Title: Study of the Effect of the Position of the Patient's Head With Brain Lesions on Cerebral Blood Flow
Brief Title: Effect of the Position of the Patient's Head
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1108183; 2011-A01565-36 (Other: ANSM)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Brain Lesion
Keywords: brain lesion; intracranial pressure; cerebral perfusion pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- position changes of head with brain lesion: patient with position changes of the head: registration of blood flow changes induced when the patient's head will be tilted at 0 ° (that is to say flat), 15 ° and 30 °.
  Interventions: Procedure: position changes of the head

INTERVENTIONS:
Procedure: position changes of the head — Registration of blood flow changes induced when the patient's head will be tilted at 0 ° (that is to say flat), 15 ° and 30 ° (the order of actions will be determined by drawing lots). The patient will remain 10 minutes in each of these positions.

SUMMARY:
The position of the head of the patient influences the cerebral venous return and cerebral perfusion pressure (CPP). In our daily practice, it is almost routine to prescribe a Trendelenburg position 30 ° in all brain-damaged patients. However, this is based only on precarious bibliographic databases. It has been shown to decrease the Intracranial Pressure (ICP) in Trendelenburg position relative to the horizontal, with varying effects on PPC. Effects on sylvian objectified by Doppler velocities and cerebral oxygenation seem unaffected by changes of position of the head of the patient. But the whole of the literature on this subject has significant bias.

DETAILED DESCRIPTION:
Registration of blood flow changes induced when the patient's head will be tilted at 0 ° (that is to say flat), 15 ° and 30 ° (the order of actions will be determined by randomization). The patient will remain 10 minutes in each of these positions and will also have a little extra blood sample of 1 ml (ie 9 samples). These measures will be carried out again the next day and then after five days to see if the results vary depending on the evolution of his condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years with:

  * A severe head injury
  * or subarachnoid hemorrhage before the 5th day of evolution
  * or spontaneous intracranial hematoma
  * or ischemic stroke
* Neurosurgical Patients after surgery
* Presenting intracranial hypertension

Exclusion Criteria:

* Hemodynamic and / or neurological instability. In the most unstable patients, care and mobilizations are reduced to a minimum.
* Craniectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with brain lesion
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation | day 1
  Value of cerebral oxygenation (Hg mm) after 5 minutes in each position

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GERGELE, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France